CLINICAL TRIAL: NCT03565939
Title: Probiotic Treatment of Ulcerative Colitis With Trichuris Suis Ova (TSO)
Acronym: PROCTO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ParaTech A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PROCTO; 2017-004772-65 (EudraCT Number)
Record Dates: First submitted 2018-05-22; First posted 2018-06-21 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis Chronic Moderate
Keywords: Ulcerative Colitis; Trichuris suis; Trichuris suis ova; Probiotic; IBD; Inflammatory bowel diseases; Anti inflammatory; Hygiene Hypothesis; Helminths; Microbiome; MAYO
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind randomised, placebo-controlled, 24 weeks, comparative, exploratory phase II proof of concept trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trichuris suis ova (TSO) (Active Comparator): 7500 TSO suspension, orally every second week for 24 weeks.
  Interventions: Biological: Trichuris suis ova
- Placebo (Placebo Comparator): Solution without TSO orally every second week for 24 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Trichuris suis ova — Eggs from the pig whipworm
  Other Names: TSO
  Arms: Trichuris suis ova (TSO)
Biological: Placebo — Solution without TSO
  Arms: Placebo

SUMMARY:
The PROCTO trial is a double-blind randomized, placebo-controlled, 24-week, comparative, exploratory phase II proof of concept trial. The trial will be conducted with 2 treatment groups as a parallel group comparison and will serve to compare a 7500 TSO regimen vs. placebo for achieving clinically meaningful responses in Ulcerative Colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Between 18 and 75 years of age
3. Established diagnosis of UC confirmed by endoscopic (sigmoidoscopy) and histological criteria, at least 3 months prior to inclusion
4. Disease extension corresponding to E2 (left side colitis) or E3 (extensive colitis) according to the Montreal Classification, i.e. at least 15 cm from anal verge, confirmed by an index sigmoidoscopy
5. Mayo-score between 6 and 10 and including 6 and 10 corresponding to moderately active disease
6. Calprotectin ≥ 250 µg/g and an endoscopic Mayo score ≥ 2
7. Negative pregnancy test in females of childbearing potential and the use of an acceptable effective method of contraception
8. No treatment or if treated with 5-Aminosalicyl acid (5-ASA): 5-ASA ≥ 8 weeks with a stable dose for at least 4 weeks both oral and rectal use
9. Tapered down from last oral steroid ≥ 4 weeks ago

Exclusion Criteria:

1. Disease extension corresponding only to E1 (proctitis), i.e. less than 15 cm from the anal verge
2. Bowel surgery, except appendectomy and removal of polyps
3. Septic complications
4. Evidence of infectious diarrhea (i.e. pathogenic bacteria or Clostridium difficile toxin in stool)
5. Abscess, perforation, active fistula or perianal lesions
6. Abnormal hepatic function (ALAT or ALP > 2.5 x ULN at screening), liver cirrhosis, or portal hypertension
7. Abnormal renal function (Creatinine > ULN) at screening
8. Any severe concomitant cardiovascular, renal, endocrine, or psychiatric disorder, which in the opinion of the investigator might have an influence on the patient's compliance or the interpretation of the results
9. Any condition associated with significant immunosuppression
10. Treatment with immunosuppressants or anti-cancer drugs, e.g., anti-TNF-α agents, anti-integrin agents, azathioprine or 6-MP, 6-thioguanine, methotrexate, tacrolimus, cyclophosphamide, or cyclosporine within the last 3 months prior to baseline
11. Treatment with systemic broad-spectrum antibiotics (e.g. metronidazole or ciprofloxacin), anti-parasitic medications, or probiotic (e.g. fecal transplantation) medication within the last 4 weeks prior to baseline, except for probiotic lactobacillus or bifidobacteria within 2 week prior to baseline (and minimum 1 week before screening visit (sampling and biopsies)).
12. Treatment with systemic glucocorticosteroid within the last 4 weeks or treatment with topical steroid within the last 2 weeks prior to baseline
13. Application of systemic non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks before baseline visit for more than 3 consecutive days, except acetylsalicylic acid ≤ 350 mg/d which is allowed
14. Immunization with live vaccines within 12 weeks prior to baseline or during the trial
15. Travelling to rural districts in countries outside of Europe, USA, Australia or Canada within the last 12 weeks prior to baseline or during trial participation. If patients travel outside of Europe, USA, Australia or Canada they must be tested negative in the standard stool tests (parasites, bacteria and virus) when they return, as at the screening visit.
16. Well-founded doubt about the patient's cooperation, (e.g., addiction to alcohol or drugs).
17. Existing or intended pregnancy or breast-feeding
18. Participation in another clinical trial within the last 60 days, simultaneous participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Remission (Full Mayo) | 24 weeks
  To achieve clinical remission defined as full Mayo score ≤ 2 at 24 weeks (long-term efficacy) (ITT, PP). The full Mayo score (range 0-12) is the sum of 4 clinical scores (stool frequency, rectal bleeding, mucosal appearance at endoscopy, physician rating of disease activity) each scored with a value 0 (normal), 1, 2, or 3 (worst).

SECONDARY OUTCOMES:
Response (Full Mayo) | 24 weeks
  To achieve reduction of full Mayo score of 4 or more steps at 24 weeks (ITT, PP, complete steroid-free)
Steroid free remission (Full Mayo) | 24 weeks
  To achieve complete steroid free clinical remission defined as full Mayo score ≤ 2 at 24 weeks (long-term efficacy) (complete steroid-free)
Endoscopic remission | 24 weeks
  To achieve endoscopic remission defined as mucosal appearance Mayo sub-score of 0 or 1 at 24 weeks (long-term efficacy) (ITT, PP, complete steroid-free)
Symptomatic remission | 12 and 24 weeks
  To achieve symptomatic remission defined as stool frequency Mayo sub-score of 0 or 1 and rectal bleeding Mayo sub-score of 0 at 12 weeks (short-term efficacy) and at 24 weeks (long-term efficacy) (ITT, PP, complete steroid-free)
Time to remission | 0-24 weeks
  To reduce time to achieve remission defined as time to achieve a pMayo score ≤ 1 and time to achieve symptomatic remission defined as stool frequency Mayo sub-score of 0 or 1 and rectal bleeding Mayo sub-score of 0 (0-24 weeks) (ITT, PP, complete steroid-free)
Time to response | 0-24 weeks
  To reduce time to achieve response defined as time to achieve reduction in pMayo score of 3 or more steps (0-24 weeks) (ITT, PP, complete steroid-free)
Disease severity | 12-24 weeks
  To decrease disease severity assessed by pMayo scores at 12 to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD, Ph.D, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No